CLINICAL TRIAL: NCT05328882
Title: Early Recurrences of Atrial Arrhythmias and Their Impact on Late Recurrence After Pulmonary Vein Isolation With Pulsed Field Ablation of Paroxysmal Atrial Fibrillation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Split, School of Medicine (Other)
Responsible Party: Principal Investigator, Lucija Lisica, Principal Investigator, University of Split, School of Medicine
Other Study IDs: 2181-147/01/06/M.S.-21-02
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Atrial Fibrillation Paroxysmal; Recurrence
Keywords: Pulsed field ablation
MeSH Terms: conditions — Atrial Fibrillation; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- ERAF after PFA: Patients with an early recurrence after pulsed field ablation of paroxysmal atrial fibrillation.
  Interventions: Other: Monitoring of paroxysmal atrial fibrillation recurrence after pulsed field catheter ablation
- no ERAF after PFA: Patients without an early recurrence after pulsed field ablation of paroxysmal atrial fibrillation.
  Interventions: Other: Monitoring of paroxysmal atrial fibrillation recurrence after pulsed field catheter ablation

INTERVENTIONS:
Other: Monitoring of paroxysmal atrial fibrillation recurrence after pulsed field catheter ablation — The implanted loop recorder will be interrogated to see how many patients had an early recurrence of AF (up to 3 months after the procedure). Then the late recurrence rate will be compared (3-12 months post-procedure) between groups with and without early recurrences.

SUMMARY:
This is a prospective, single-arm study conducted in University Hospital of Split, Department of Cardiology. Patients treated with PFA for symptomatic paroxysmal atrial fibrillation will be asked to participate in the study. An implantable loop recorder (ILR) will be placed immediately after the PFA procedure for rhythm monitoring. Early recurrences will be subsequently divided into very early recurrences (up to 1 month post-procedure) and early recurrences (1-3 months post-procedure). Late recurrences will be defined as those 3 to 12 months post-procedure. Patients will be monitored routinely through follow up visits during which ILR will be interrogated and eventual symptoms will be assessed. Follow-up visits will be scheduled 1, 3, 6, 12 months post-procedure. Median follow-up will be 12 months. Data for the study will be obtained from a loop monitor to assess the arrhythmia burden during follow-up visits in the University Hospital of Split Arrhythmia Clinic.

DETAILED DESCRIPTION:
This is a prospective, single-arm study conducted in the University Hospital of Split, Department of Cardiology. Patients treated with PFA for symptomatic paroxysmal atrial fibrillation will be asked to participate in the study. An implantable loop recorder (ILR) will be placed immediately after the PFA procedure for rhythm monitoring. Early recurrences will be subsequently divided into very early recurrences (up to 1-month post-procedure) and early recurrences (1-3 months post-procedure). Late recurrences will be defined as those 3 to 12 months post-procedure. Patients will be monitored routinely through follow-up visits during which ILR will be interrogated and eventual symptoms will be assessed. Follow-up visits will be scheduled 1, 3, 6, and 12 months post-procedure. The median follow-up will be 12 months. Data for the study will be obtained from a loop monitor to assess the arrhythmia burden during follow-up visits in the University Hospital of Split Arrhythmia Clinic.

For PVI, the "single-shot" multielectrode PFA catheter will be used. This catheter consists of 5 splines, with 4 electrodes per spline and 1 electrode available for intracardiac electrogram recording or 3-dimensional electroanatomic visualization. When used in conjunction with the PFA generator, an electric field is created that ablates tissue using irreversible electroporation. The catheter shape is changed through the manipulation of a slider mechanism on the handle of the catheter. The diameter of the catheter is measured in the fully deployed "flower" configuration and is available in 2 sizes (31 or 35 mm). Energy is delivered through all of the electrodes in a proprietary sequence.

All patients will be asked to provide written informed consent for their respective protocol before undergoing the study.

All procedures will be performed with conscious sedation and propofol bolus synchronized to sets of PFA applications. The procedures will be performed with uninterrupted oral anticoagulation, and left atrial thrombus will be excluded either through pre-procedure CT or intracardiac echocardiography (ICE) (AcuNav, Siemens, Munich, Germany) at the time of the procedure. Pre- and post-ablation diaphragm motion will be evaluated to observe changes in phrenic nerve function during the procedure. Esophageal temperature monitoring will not be utilized due to the nonthermal nature of PFA.

A single transseptal puncture will be performed with an 8.5-F sheath and exchanged for the 13-F PFA sheath in the left atrium, or a transseptal puncture will be performed directly with the PFA sheath. Intravenous heparin will be administered as boluses and continuous infusions to obtain an activated clotting time ≥300 s prior to ablation and throughout the procedure. A 0.035-inch, 180-cm extra-stiff, straight guidewire will be used to cannulate each vein over which the multielectrode PFA catheter will be deployed into the desired shape and advanced into position at the antrum of each vein. The antral level of catheter positioning will be monitored with ICE imaging and fluoroscopy. Patients with left common PV anatomy will receive therapy at the level of the common antrum with 2 sets of therapy delivered, 1 with the guidewire in a superior branch and 1 with the guidewire in an inferior branch.

Acute isolation of the treated vein will be determined by the mapping electrodes on each spline of the PFA catheter. Once all veins have been treated, a 3-dimensional electroanatomic voltage map will be created to confirm PV isolation and visualize the level of isolation of each lesion set. Entrance or exit block will be confirmed following a 20-min wait period after the last PFA application was delivered with a circular mapping catheter (Lasso, Biosense Webster, Irvine, California).

All patients will be implanted with an ILR (Medtronic Reveal LINQTM; Medtronic, Minneapolis, MN). After ablation procedure, the ILR will be inserted subcutaneously in the left fourth intercostal space. The procedure itself takes up to 15 minutes and local anesthetic will be administered prior to the implantation. The antiarrhythmic drugs, except beta-blocker, will be routinely discontinued.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Index PFA procedure after one failed or intolerant group I or III of the antiarrhythmic drug in patients with symptomatic paroxysmal AF (AF with self-terminating episodes lasting no longer than 7 continuous days)
* Willing and able to provide informed consent.

Exclusion Criteria:

* Any known contraindication to AF ablation or anticoagulation.
* History of previous left atrial ablation or surgical treatment.
* Secondary AF due to reversible or non-cardiac cause such as thyroid disease and electrolyte imbalance.
* Asymptomatic AF patients, persistent AF, permanent AF patients.
* History of clotting or bleeding disease or cryoglobulinemia.
* Pregnant or lactating.
* Other conditions that may make the patient a poor candidate for procedure such as mental illness, terminal illness, vulnerable patient population.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic paroxysmal atrial fibrillation after at least one failed or intolerant group I or III of antiarrhythmic drug that are eligible for PFA and are willing and able to provide informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-11-17 (Actual); Primary Completion 2024-05-17 (Estimated); Study Completion 2024-05-17 (Estimated)

PRIMARY OUTCOMES:
Number of participants with AF recurrence 3-12 months post-procedure | 12 months
  Number of participants with AF recurrence 3-12 months post-procedure (AF burden defined by loop recorder findings)

SECONDARY OUTCOMES:
Adverse event rate | 12 months
  Adverse event rate defined as any untoward medical occurrence, unintended disease or injury related to all aspects of the ablation procedure (death, air embolism, myocardial infarction, stroke, esophageal injury, PV stenosis, puncture site hematoma, vascular lesions).
Number of patients with very early AF recurrence (within 1 month post procedure) | 12 months
  Number of patients with very early AF recurrence (within 1 month post procedure)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Center Split, Split, Split-Dalmatia County, Croatia

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become available immediately after the publication of the study.
Access Criteria: The plan will be shared with other researchers who wish to replicate the study or study the protocol in detail.

REFERENCES:
- [Background] Hindricks G, Potpara T, Dagres N, Arbelo E, Bax JJ, Blomstrom-Lundqvist C, Boriani G, Castella M, Dan GA, Dilaveris PE, Fauchier L, Filippatos G, Kalman JM, La Meir M, Lane DA, Lebeau JP, Lettino M, Lip GYH, Pinto FJ, Thomas GN, Valgimigli M, Van Gelder IC, Van Putte BP, Watkins CL; ESC Scientific Document Group. 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS): The Task Force for the diagnosis and management of atrial fibrillation of the European Society of Cardiology (ESC) Developed with the special contribution of the European Heart Rhythm Association (EHRA) of the ESC. Eur Heart J. 2021 Feb 1;42(5):373-498. doi: 10.1093/eurheartj/ehaa612. No abstract available. PMID 32860505
- [Background] Tanno K, Kobayashi Y, Kurano K, Kikushima S, Yazawa T, Baba T, Inoue S, Mukai H, Katagiri T. Histopathology of canine hearts subjected to catheter ablation using radiofrequency energy. Jpn Circ J. 1994 Feb;58(2):123-35. doi: 10.1253/jcj.58.123. PMID 8196154
- [Background] Grubman E, Pavri BB, Lyle S, Reynolds C, Denofrio D, Kocovic DZ. Histopathologic effects of radiofrequency catheter ablation in previously infarcted human myocardium. J Cardiovasc Electrophysiol. 1999 Mar;10(3):336-42. doi: 10.1111/j.1540-8167.1999.tb00680.x. PMID 10210495
- [Background] Malmborg H, Christersson C, Lonnerholm S, Blomstrom-Lundqvist C. Comparison of effects on coagulation and inflammatory markers using a duty-cycled bipolar and unipolar radiofrequency pulmonary vein ablation catheter vs. a cryoballoon catheter for pulmonary vein isolation. Europace. 2013 Jun;15(6):798-804. doi: 10.1093/europace/eus411. Epub 2013 Jan 29. PMID 23362019
- [Background] Calkins H, Hindricks G, Cappato R, Kim YH, Saad EB, Aguinaga L, Akar JG, Badhwar V, Brugada J, Camm J, Chen PS, Chen SA, Chung MK, Cosedis Nielsen J, Curtis AB, Davies DW, Day JD, d'Avila A, Natasja de Groot NMS, Di Biase L, Duytschaever M, Edgerton JR, Ellenbogen KA, Ellinor PT, Ernst S, Fenelon G, Gerstenfeld EP, Haines DE, Haissaguerre M, Helm RH, Hylek E, Jackman WM, Jalife J, Kalman JM, Kautzner J, Kottkamp H, Kuck KH, Kumagai K, Lee R, Lewalter T, Lindsay BD, Macle L, Mansour M, Marchlinski FE, Michaud GF, Nakagawa H, Natale A, Nattel S, Okumura K, Packer D, Pokushalov E, Reynolds MR, Sanders P, Scanavacca M, Schilling R, Tondo C, Tsao HM, Verma A, Wilber DJ, Yamane T; Document Reviewers:. 2017 HRS/EHRA/ECAS/APHRS/SOLAECE expert consensus statement on catheter and surgical ablation of atrial fibrillation. Europace. 2018 Jan 1;20(1):e1-e160. doi: 10.1093/europace/eux274. No abstract available. PMID 29016840
- [Background] Willems S, Khairy P, Andrade JG, Hoffmann BA, Levesque S, Verma A, Weerasooriya R, Novak P, Arentz T, Deisenhofer I, Rostock T, Steven D, Rivard L, Guerra PG, Dyrda K, Mondesert B, Dubuc M, Thibault B, Talajic M, Roy D, Nattel S, Macle L; ADVICE Trial Investigators*. Redefining the Blanking Period After Catheter Ablation for Paroxysmal Atrial Fibrillation: Insights From the ADVICE (Adenosine Following Pulmonary Vein Isolation to Target Dormant Conduction Elimination) Trial. Circ Arrhythm Electrophysiol. 2016 Aug;9(8):e003909. doi: 10.1161/CIRCEP.115.003909. PMID 27516462
- [Background] Mariani MA, Pozzoli A, Maat G, Alfieri OR, Benussi S. What Does The Blanking Period Blank? J Atr Fibrillation. 2015 Dec 31;8(4):1268. doi: 10.4022/jafib.1268. eCollection 2015 Dec. PMID 27957225
- [Background] Reddy VY, Anic A, Koruth J, Petru J, Funasako M, Minami K, Breskovic T, Sikiric I, Dukkipati SR, Kawamura I, Neuzil P. Pulsed Field Ablation in Patients With Persistent Atrial Fibrillation. J Am Coll Cardiol. 2020 Sep 1;76(9):1068-1080. doi: 10.1016/j.jacc.2020.07.007. PMID 32854842
- [Background] Calkins H, Gache L, Frame D, Boo LM, Ghaly N, Schilling R, Deering T, Duytschaever M, Packer DL. Predictive value of atrial fibrillation during the postradiofrequency ablation blanking period. Heart Rhythm. 2021 Mar;18(3):366-373. doi: 10.1016/j.hrthm.2020.11.020. Epub 2020 Nov 24. PMID 33242668
- [Background] Reddy VY, Dukkipati SR, Neuzil P, Anic A, Petru J, Funasako M, Cochet H, Minami K, Breskovic T, Sikiric I, Sediva L, Chovanec M, Koruth J, Jais P. Pulsed Field Ablation of Paroxysmal Atrial Fibrillation: 1-Year Outcomes of IMPULSE, PEFCAT, and PEFCAT II. JACC Clin Electrophysiol. 2021 May;7(5):614-627. doi: 10.1016/j.jacep.2021.02.014. Epub 2021 Apr 28. PMID 33933412
- [Background] Reddy VY, Neuzil P, Koruth JS, Petru J, Funosako M, Cochet H, Sediva L, Chovanec M, Dukkipati SR, Jais P. Pulsed Field Ablation for Pulmonary Vein Isolation in Atrial Fibrillation. J Am Coll Cardiol. 2019 Jul 23;74(3):315-326. doi: 10.1016/j.jacc.2019.04.021. Epub 2019 May 11. PMID 31085321
- [Background] Kawamura I, Neuzil P, Shivamurthy P, Petru J, Funasako M, Minami K, Kuroki K, Dukkipati SR, Koruth JS, Reddy VY. Does pulsed field ablation regress over time? A quantitative temporal analysis of pulmonary vein isolation. Heart Rhythm. 2021 Jun;18(6):878-884. doi: 10.1016/j.hrthm.2021.02.020. Epub 2021 Feb 27. PMID 33647464
- [Background] Stewart MT, Haines DE, Verma A, Kirchhof N, Barka N, Grassl E, Howard B. Intracardiac pulsed field ablation: Proof of feasibility in a chronic porcine model. Heart Rhythm. 2019 May;16(5):754-764. doi: 10.1016/j.hrthm.2018.10.030. Epub 2018 Oct 30. PMID 30385383
- [Background] Kim YG, Boo KY, Choi JI, Choi YY, Choi HY, Roh SY, Shim J, Kim JS, Kim YH. Early Recurrence Is Reliable Predictor of Late Recurrence After Radiofrequency Catheter Ablation of Atrial Fibrillation. JACC Clin Electrophysiol. 2021 Mar;7(3):343-351. doi: 10.1016/j.jacep.2020.09.029. Epub 2021 Jan 27. PMID 33516711